CLINICAL TRIAL: NCT03612414
Title: Effetti Sulla Salivazione a Seguito Della Somministrazione di un Integratore Alimentare (Aqualief®) a Base di Carnosina ed Hibiscus Nei Soggetti Xerostomici: Studio Multicentrico, Randomizzato, in Doppio Cieco, Controllato Verso Placebo
Brief Title: Efficacy of a Dietary Supplement (Aqualief®) in Xerostomic Patients
Acronym: Aqualief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Prof. Luca Levrini, Director of the Department of Surgery and Medicine, Dental Hygiene School, Research Centre Cranio Facial Disease and Medicine, University of Insubria, Varese Italy, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Prot.49 May 31st, 2016
Record Dates: First submitted 2018-07-04; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland; pH; Saliva; Quality of Life
Keywords: xerostomia; pH; Carnosine; karkadé; Aqualief; Mucoadhesive
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled clinical study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqualief® tablets (Experimental): 400 mg mucoadhesive tablets; three times per day just
  Interventions: Dietary Supplement: Aqualief
- Placebo tablets (Placebo Comparator): 400 mg mucoadhesive placebo tablets, three times per day just
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aqualief — Three tablets/day
  Arms: Aqualief® tablets
Dietary Supplement: Placebo — Three tablets/day
  Arms: Placebo tablets

SUMMARY:
Xerostomia is defined as the subjective complaint of dry mouth. Symptoms of dry mouth may range from mild oral discomfort to significant oral disease that can compromise patients' health, dietary intake and quality of life. Xerostomia is accompanied by numerous signs and symptoms mainly in the mucous membranes, lips, tongue, salivary glands and teeth.

This study was designed to verify efficacy and safety of a novel dietary supplement (Aqualief),designed with the aim of stabilizing the saliva flux and pH at a neutral level and to improve the acid buffering capacity of saliva.

DETAILED DESCRIPTION:
Sixty patients with xerostomia (grade 1-2 according to RTOG/EORTC) from different etiologies were recruited at the Clinica Odontoiatrica dell'Università degli studi dell'Insubria (Varese, Italy). Exclusion criteria were subjects under treatment using drugs to treat hyposalivation (e.g. pilocarpine) and xerostomia grade ≥ 3. Patients with severe hyposalivation were excluded (saliva flow rate at baseline <0.1 ml min-1) due to their inability to dissolve the tablet formulation.

Written informed consent was received from all patients before study initiation. The study was conducted in accordance with the principles laid out by the Declaration of Helsinki 1964 and its subsequent amendments and with the International Committee on Harmonization Guidelines for Good Clinical Practice and in compliance with local ethical and legal requirements. The study was approved by the ethics committee at the participating site.

The study was a prospective, randomized, double-blind, placebo-controlled trial undertaken at the Clinica Odontoiatrica dell'Università degli Studi dell'Insubria (Varese, Italy). Eligible patients who had developed xerostomia RTOG/EORTC grade 1-2 were randomized in a 1:1 ratio, with one group receiving three Aqualief tablets (after meals: breakfast, lunch, dinner) daily for 6 days. The second group received a placebo tablet given with the same regimen. The primary objective of the study was to assess the safety and efficacy of Aqualief in stabilizing the saliva pH at a neutral level compared with placebo. The secondary objective was to determine whether Aqualief induced an increase of unstimulated or stimulated saliva and in ameliorating the symptoms related to oral dryness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sex
* Age ≥ a 18 years
* Able to understand and sign the Informed Consent, and fill in the patient's diary
* Subjects suffering from Xerosotmia Grade 1-2 (according to RTOG/EORTC scale)
* Sjögren Sindrome
* Lambert-Eaton Sindrome
* Diabetes mellitus and low metabolic control
* Anxiety
* Alcool abuse
* Salivary glands trauma
* Radio and Chemotherapy for head & neck cancer
* Methamphetamine, cannabis, heroin abuse
* Xerostomia caused by (single and concomitant, i.e. Anti-depressive and anxyolitic drugs; Antihistaminic drugs; Decongestive drugs; Antihypertensive drugs; Muscle relaxants; Urinary incontinence drugs; Drugs for Parkinson treatment)
* Subjects affected by paradental pathology diagnosed according to AAOP criteria, PSR 2-3

Exclusion Criteria:

* Contraindication and/or Hypersensitivity to product's components, and in particular carnosine and Hibiscus
* Subjects that are under treatment with products or drugs ( ie pilocarpin) for hypofunctionality of salivary glands
* Subjects with total ablation of salivary glands caused by chemo or radiotherapy
* Use of experimental drugs during 30 days before the enrolment or during the study
* Conditions that can interfere with the study
* Xerostomia grade 3 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Effect of Aqualief on salivation | Change from baseline to 6 days of treatment
  Changes in saliva production is measured (ml)

SECONDARY OUTCOMES:
Safety of Aqualief | Occurrence of Adverse Events over the 6 days of treatment
  Incidence of Treatment-Emergent Adverse Events
Effect of Aqualief on dry mouth symptoms | Change from baseline to 6 days of treatment
  Evaluate the effect of treatments dry mouth symptoms trough Dry Mouth Questionnaire (Thomson Questionnaire)
Effect of Aqualief on the pH of saliva | Change from baseline to 6 days of treatment
  Changes of saliva pH is measured

CONTACTS AND LOCATIONS:
Overall Officials: Luca Levrini, Prfo. MD., Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Università degli Studi dell'Insubria, Varese, Italy